CLINICAL TRIAL: NCT04964375
Title: A Phase 1, Open-Label Study of ABSK043 to Assess Safety, Tolerability, and Pharmacokinetics in Patients With Advanced Solid Tumor
Brief Title: A Study to Assess Safety, Tolerability, and Pharmacokinetics of ABSK043 in Patients With Advanced Solid Tumor
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abbisko Therapeutics Co, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ABSK043-101
Record Dates: First submitted 2021-06-24; First posted 2021-07-16 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2021-07

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ABSK043 (Experimental): Dose escalation of oral ABSK043 with a starting dose of 200mg once daily will be guided by"BOIN" escalation rules based on safety data until an MTD has been identified or a RDE. For each dose,In the escalation part, sequential cohorts of patients will receive an oral dose of ABSK043 in repeated 28-day cycles. Starting dose level will be 200 mg QD. Cohort 3 on 800mg will be switched to 400mg BID.Then, patients will continuously receive ABSK043 （total daily dose） in repeated 28-day cycles.For the Dose Expansion Phase, patients will each receive orally administered doses of ABSK043 at the RDE in repeated 28-day cycles.
  Interventions: Drug: ABSK043 oral capsule

INTERVENTIONS:
Drug: ABSK043 oral capsule — ABSK043 is a novel, oral small molecule inhibitor of PD-L1

SUMMARY:
This is a Phase 1, Open-Label Study of ABSK043 to Assess Safety, Tolerability, and Pharmacokinetics in Patients with Advanced Solid Tumor.

Preliminary antitumor activity will also be assessed. Investigate the pharmacodynamics (PD) effects and Investigate the metabolites of oral ABSK043

DETAILED DESCRIPTION:
The study will start with a dose escalation part of single-agent ABSK043 administered in repeated 28-day cycles in patients with advanced solid for safety and tolerability. The expansion part of oral ABSK043 at recommended dose of expansion (RDE) will be followed for further evaluating safety and tolerability among selected tumor types. Preliminary antitumor activity will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should understand, sign, and date the written voluntary informed consent form prior to screening.
2. Male or female aged 18 years or older (or other age range required by local regulations or IRB).
3. For Escalation part: patients must have histologically confirmed solid tumors that have progressed on or intolerance to standard therapy or whom no standard therapy exists or whom refuse to receive standard therapy；

For Expansion Part:

1. Melanoma cohort: Patients must have histologically confirmed melanoma that have have progressed on or intolerance to standard therapy(including immune-checkpoint inhibitors) or whom no standard therapy exists or whom refuses to receive standard therapy
2. MSI-H/dMMR cohort: Patients must have histologically confirmed solid tumors harboring MSI-H or dMMR that have progressed on or intolerance to standard therapy or whom no standard therapy exists or whom refuses to receive standard therapy.
3. Patients must have at least one measurable target lesion according to RECIST 1.1.
4. Patients are willing to receive biopsy. 4. ECOG performance status 0 or 1 5. Life expectancy ≥3 months 6. Adequate organ function and bone marrow function as indicated by the following screening assessments performed within 14 days prior to the first dose of study drug:

   1. Absolute neutrophil count (ANC) ≥1.5×109/L
   2. Platelet count (PLT) ≥75×109/L without transfusions within 14 days before 1st dose
   3. Hemoglobin (Hb) ≥90 g/L
   4. Total bilirubin (TBIL) ≤1.5×ULN
   5. Aspartate transaminase (AST)/alanine transaminase (ALT), ≤3×ULN (≤5 × ULN in the presence of hepatic metastases).
   6. Serum creatinine (Cr) of ≤1.5×ULN for the reference laboratory or creatinine clearance (Crcl) ≥50 mL/min based either on urine collection or Cockcroft-Gault estimation

Exclusion Criteria:

1. Known allergy or hypersensitivity to any component of the investigational product.
2. For expansion part MSI-H or dMMR cohort only: previously treated with PD-(L)1 pathway inhibitors (including monoclonal antibody and small molecular agents).
3. History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis, etc.
4. History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan, history of radiation pneumonitis in the radiation field (fibrosis) is permitted.
5. For expansion part only: Has a known additional malignancy that is progressing or required active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy, or other in situ cancers.
6. Inability to take oral medication or significant nausea and vomiting, malabsorption, external biliary shunt, or significant bowel resection that would preclude adequate absorption of oral medication.
7. Previous anti-cancer therapy, including chemotherapy (chemotherapy with nitrosourea or mitomycin should be 6 weeks prior to initiation of study treatment), radiotherapy, molecular targeted therapy or other investigational drugs received in previous clinical trial ≤4 weeks; endocrine therapy ≤2 weeks or ≤5-half-life (whichever is shorter) prior to initiation of study treatment.
8. Major surgery within 4 weeks of the first dose of study drug and all surgical wounds must be healed and free of infection or dehiscence.
9. Vaccination with a live, attenuated vaccine within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivate vaccines (e.g., COVID-19 vaccines, inactivated influenza vaccines).
10. Prior toxicities from chemotherapy, radiotherapy, and other anti-cancer therapies, including immunotherapy that have not regressed to Grade ≤1 severity (CTCAE v5.0) with the exception of alopecia, vitiligo or event(s) that is considered non-clinical meaningful by the Investigator.
11. History of Grade ≥3 immune-related adverse event(s) occurred in previous treatment.
12. Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 2 weeks prior to randomization, or anticipated requirement for systemic immunosuppressive medications during the trial (patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study; patients with a history of allergic reaction to IV contrast requiring steroid pre-treatment should have baseline and subsequent tumor assessments performed using MRI; the use of inhaled corticosteroids for chronic obstructive pulmonary disease, mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension, and low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed.
13. For expansion part only: last treatment with therapeutic oral or intravenous antibiotics within 2 weeks prior to first dose of study treatment.
14. Concomitant use of the drugs/remedies that may cause pharmacokinetic drug-drug interactions; Consumption of grapefruit juice, grapefruit hybrids, pomegranates, starfruit, pomelos, Seville oranges or juice or products within 7 days prior to the first dose of study medication (for Escalation Part only).
15. Active central nervous system (CNS) metastases including cerebral edema, system hormone treatment, disease progression due to intracranial lesions, leptomeningeal metastasis, and other clinical symptoms related to CNS metastases (if stable disease>8 weeks after treatment and free from glucocorticoids can be enrolled).
16. Impaired cardiac function or clinically significant cardiac disease, including any one of the following:

    * New York Heart Association class III or IV heart disease, active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiacarrhythmia requiring therapy, uncontrolled hypertension or congestive heart failure.
    * Baseline prolongation of the rate-corrected QT interval based on repeated demonstration of QTcF >480 ms or history of long QT interval corrected (QTc) syndrome (Note: QTc interval corrected by Fridericia's formula). Left ventricular ejection fraction (LVEF) <50% or below the lower limit of normal(whichever is higher)
17. Known human immunodeficiency virus or active hepatitis B, or active hepatitis C infection or active tuberculosis. Positive tests for hepatitis B virus surface antigen (HBsAg), or antibody to hepatitis B core Ag or hepatitis C RNA in serum. (subjects with history of hepatitis C infection but negative hepatitis C virus polymerase chain reaction (PCR) test and subjects with hepatitis B with positive hepatitis B surface antibody are allowed)
18. Patients with refractory/uncontrolled ascites or pleural effusion. Patients with indwelling catheters are allowed.
19. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test within 7 days prior to the start of study drug.
20. Non-surgically sterilized male or female patients of childbearing potential must agree to use effective methods of birth control during the study and for up to 6 months after the last dose of study drug.
21. Sexually active males unless they use a condom during intercourse while taking drug and for 5 compound half-lives plus 60 days after stopping study drug and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
22. Any other clinically significant comorbidities, such as uncontrolled pulmonary disease, active infection, or any other condition, which in the judgment of the Investigator, could compromise compliance with the protocol, interfere with the interpretation of study results, or predispose the patient to safety risks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2022-10-23 (Estimated); Study Completion 2023-03-23 (Estimated)

PRIMARY OUTCOMES:
DLT | At the end of Cycle 1 (each cycle is 28 days)
  dose-limiting toxicity
Incidence and Severity of AEs | Through study completion, an average of 6 months
  Adverse events (AEs), adverse events of special interest (AESIs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
PFS | throughout study completion, on average of half year
  Progression-Free Survival
DCR | throughout study completion, on average of half year
  Disease control rate up to 24 weeks
DOR | throughout study completion, on average of half year
  Duration of response
Cmax | at the end of Cycle 1 Day15 (each cycle is 28 days)
  maximun observed concentration
Tmax | at the end of Cycle 1 Day15 (each cycle is 28 days)
  time to maximum observed concentration
AUC | at the end of Cycle 1 Day15 (each cycle is 28 days)
  area under the concentration-time curve
t1/2 | at the end of Cycle 1 Day15 (each cycle is 28 days)
  half-life
Vz/F | at the end of Cycle 1 Day15 (each cycle is 28 days)
  apparent volume of distribution
CL/F | at the end of Cycle 1 Day15 (each cycle is 28 days)
  apparent oral clearance
Css_max | at the end of Cycle 1 Day15 (each cycle is 28 days)
  maximun observed concentration of steady-state
Css_min | at the end of Cycle 1 Day15 (each cycle is 28 days)
  minimum observed concentration of steady-state
AUCss | at the end of Cycle 1 Day15 (each cycle is 28 days)
  area under the concentration-time curve of steady-state
Rac | at the end of Cycle 1 Day15 (each cycle is 28 days)
  accumulation rate
ORR | throughout study completion, on average of half year
  Overall response rate

OTHER OUTCOMES:
surface PD-L1 expression | Time Frame:at the end of Cycle 1 Day15 (each cycle is 28 days)
  Programmed death-ligand 1
metabolites of ABSK043 | Time Frame: at the end of Cycle 1 Day15 (each cycle is 28 days)
  any major active metabolites
soluble PD-L1, | Time Frame:at the end of Cycle 1 Day15 (each cycle is 28 days)
  Programmed death-ligand 1

CONTACTS AND LOCATIONS:
Overall Officials: Jermaine Coward, Principal Investigator — Icon Cancer Centre South Brisbane
Locations (3):
- Australia (3):
  - Icon Cancer Centre South Brisbane, Brisbane, Queensland
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Sydney South West Private Hospital, Liverpool